CLINICAL TRIAL: NCT00279838
Title: Computer Assisted Navigation in Total Knee Arthroplasty
Brief Title: Computer Assisted Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: DePuy Orthopaedics (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 957-04
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Procedure: Computer Assisted Navigation Knee Replacement

SUMMARY:
The purpose of this study is to determine whether intraoperative computer-assisted navigation improves prosthetic implant positioning as compared to conventional intraoperatve instrumentation in Total Knee Arthroplasty (TKA).

DETAILED DESCRIPTION:
Primary data to be obtained is to determine whether mechanical axis of the limb malignment differs between patients whom have computer-assisted TKA and those treated with conventional intraoperative instrumentation.

Three months after surgery follow-up radiographic data will provide evidence on the initial implant position as determined with a series of x-rays including: full length standing, standard AP weight bearing, lateral, patellar, kneelingfilm views and CT evaluation. In addition, a correlation betweeen the CT measures and the kneeling x-ray can be performed at this time. Clinical (Knee Scale Society, WOMAC, and SF-36) data will also be obtained at the three month interval.

ELIGIBILITY:
Study participants must:

1. Be over 18 years of age.
2. Require a TKA and is considered by the investigator to be a suitable candidate for the specific knee prosthesis identified in protocol.
3. The subject has given consent to the transfer of his/her information to the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To determine whether mechanical axis of the limb malalignment differs between patients whom have computer-assisted TKA and those treated with conventional intraoperative instrumentation

SECONDARY OUTCOMES:
To compare the frontal alignment of the femoral and tibial components from full length standing radiographs
To compare sagittal alignment of the femoral and tibial components from lateral radiographs
To compare the rotation of the femoral and tibial components from CT Scan.

CONTACTS AND LOCATIONS:
Overall Officials: Mary I. O'Connor, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States